CLINICAL TRIAL: NCT02814162
Title: Predictive Values of Serum Adiponectin Levels in Aneurysmal Subarachnoid Hemorrhage.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKSAH
Record Dates: First submitted 2016-05-02; First posted 2016-06-27 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Subarachnoid Hemorrhage, Aneurysmal; Predictive; Adiponectin
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the predictive value of serum adiponectin levels in aneurysmal subarachnoid hemorrhage patients.

DETAILED DESCRIPTION:
Adiponectin (APN) is an abundant protein hormone derived from adipose tissue. It has been suggested to exert anti-inflammatory, antiatherogenic, and vascular protective. Subarachnoid hemorrhage (SAH) comprises about 5% of all strokes with high mortality and permanent disability rates. Although many patients survive from the initial hemorrhage or rebleeding, they suffered from long-term delayed neurological deficits (DNDs), including stroke, delayed cerebral ischemia, cognitive and neuropsychological abnormalities that seriously impact overall function and quality of life. Ruptured cerebral aneurysms are the most common cause of SAH. There is growing evidence supporting APN act as a predictive factor for SAH. The observational study will focus on the predictive value of serum adiponectin levels in aneurysmal subarachnoid hemorrhage (aSAH).

ELIGIBILITY:
Inclusion Criteria:

* Age>18yrs and age<90yrs
* It shows subarachnoid hemorrhage (SAH) based on computed tomography (CT) scan on admission
* Aneurysmal subarachnoid hemorrhage confirmed by computed tomography angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography (DSA)
* SAH grade is assessed by Hunt & Hess classification
* Informed consented

Exclusion Criteria:

* Traumatic subarachnoid hemorrhage
* Patients with cerebral herniation or highly possible to occur within 2 days from SAH
* Length of hospital stay is expected to be less than 5 days
* Duration from onset to admission is more than 48 hours
* Disturbance of communication or poor compliance to blood collection, imaging examination and follow-up

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aneurysmal subarachnoid hemorrhage who are hospitalized within 24 hours from onset.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of cerebral vasospasm and delayed cerebral ischemia | 30 days post SAH
  Proved by clinical and radiologic evidence

SECONDARY OUTCOMES:
Death | 30 days post SAH
National institutes of health stroke scale (NIHSS) score | On discharge or 14 days (whichever occurs first) and 30 days post SAH
  Assessing by senior neurosurgeons
Modified Rankin scale (mRS) | 30 days and 90days post SAH
  By phone call following-up

CONTACTS AND LOCATIONS:
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thundyil J, Tang SC, Okun E, Shah K, Karamyan VT, Li YI, Woodruff TM, Taylor SM, Jo DG, Mattson MP, Arumugam TV. Evidence that adiponectin receptor 1 activation exacerbates ischemic neuronal death. Exp Transl Stroke Med. 2010 Aug 11;2(1):15. doi: 10.1186/2040-7378-2-15. PMID 20701790
- [Background] Osuka K, Watanabe Y, Yasuda M, Takayasu M. Adiponectin activates endothelial nitric oxide synthase through AMPK signaling after subarachnoid hemorrhage. Neurosci Lett. 2012 Apr 11;514(1):2-5. doi: 10.1016/j.neulet.2011.12.041. Epub 2012 Jan 3. PMID 22230897
- [Background] Psilopanagioti A, Papadaki H, Kranioti EF, Alexandrides TK, Varakis JN. Expression of adiponectin and adiponectin receptors in human pituitary gland and brain. Neuroendocrinology. 2009;89(1):38-47. doi: 10.1159/000151396. Epub 2008 Aug 13. PMID 18698133
- [Background] Kos K, Harte AL, da Silva NF, Tonchev A, Chaldakov G, James S, Snead DR, Hoggart B, O'Hare JP, McTernan PG, Kumar S. Adiponectin and resistin in human cerebrospinal fluid and expression of adiponectin receptors in the human hypothalamus. J Clin Endocrinol Metab. 2007 Mar;92(3):1129-36. doi: 10.1210/jc.2006-1841. Epub 2007 Jan 9. PMID 17213280
- [Background] Kusminski CM, McTernan PG, Schraw T, Kos K, O'Hare JP, Ahima R, Kumar S, Scherer PE. Adiponectin complexes in human cerebrospinal fluid: distinct complex distribution from serum. Diabetologia. 2007 Mar;50(3):634-42. doi: 10.1007/s00125-006-0577-9. Epub 2007 Jan 23. PMID 17242917
- [Background] Efstathiou SP, Tsioulos DI, Tsiakou AG, Gratsias YE, Pefanis AV, Mountokalakis TD. Plasma adiponectin levels and five-year survival after first-ever ischemic stroke. Stroke. 2005 Sep;36(9):1915-9. doi: 10.1161/01.STR.0000177874.29849.f0. Epub 2005 Aug 18. PMID 16109902
- [Background] Takeuchi S, Wada K, Otani N, Osada H, Nagatani K, Mori K. Temporal profile of plasma adiponectin level and delayed cerebral ischemia in patients with subarachnoid hemorrhage. J Clin Neurosci. 2014 Jun;21(6):1007-10. doi: 10.1016/j.jocn.2013.10.020. Epub 2013 Dec 22. PMID 24594449